CLINICAL TRIAL: NCT05057728
Title: Effectiveness and Mechanisms of a Multi-Focused Prevention Program Combining Face to Face With Technology-Assisted Intervention for Preschoolers' Behavior Problems
Brief Title: Effectiveness of the Social-Emotional Prevention Program Enhanced Version
Acronym: SEP+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Catrinel Alice Stefan, Lecturer, PhD, Babes-Bolyai University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PN-III-P1-1.1-TE-2019-0226
Record Dates: First submitted 2021-09-13; First posted 2021-09-27 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Child Behavior Problem
Keywords: social-emotional competence; externalizing problems; internalizing problems; parenting practices; parent stress

STUDY DESIGN:
Intervention Model Description: Participants in the current study will be assigned to either: 1) the intervention condition, which will receive the SEP+; or 2) the wait-list control group. A partially-randomized controlled trial (RCT) will be employed, in which schools will be randomly assigned to either the intervention or control group, so that all classrooms within a school will either receive the SEP+ or not. This was done in order to prevent contamination effects, which are more likely to occur when classrooms from the same school participate in the intervention and others do not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (SEP+) (Experimental): SEP+ is designed as a multi-focused (child, teacher, parent) school-based intervention, which can be employed as either a universal (i.e. targeting all children) or an indicated prevention program (i.e. targeting specifically children at risk for behavior problems). The SEP+ intervention comprises three types of intervention: 1) the classroom-based intervention in the form of a curriculum of 43 activities (2-3 activities/week) delivered over 4-months aimed at developing social-emotional skills; 2) a 6-sessions (2-2.5h/session) teacher training focused on increasing the use of positive discipline strategies and developing coaching skills for supporting children's social-emotional learning; and 3) a 6 sessions parent training (1.5.-2h/session) aiming to teach ways to manage parenting stress, to increase parent-child quality time, support children's emotion regulation and problem-solving, as well as increase positive discipline strategies.
  Interventions: Behavioral: Social-Emotional Prevention Program enhanced version

INTERVENTIONS:
Behavioral: Social-Emotional Prevention Program enhanced version — The intervention is provided for all children for whom parental consent is obtained. The intervention includes a classroom curriculum, teacher training and parent training.
  Other Names: SEP+

SUMMARY:
The current study is intended to investigate the effectiveness of the Social-Emotional Prevention Program enhanced version (SEP+) for increasing preschoolers' social-emotional competencies and reducing their risk for behavior problems.

Hypotheses for the current study are put forward for child- and parent-related outcomes. First, for the SEP+ effects for child-related outcomes, the investigators expect that: 1) intervention group children will be rated significantly higher on measures of social-emotional competencies (social skills and positive emotion regulation strategies (ER)) compared to children from the wait-list control group (primary outcomes); and 2) children assigned to the intervention will be rated significantly lower on externalizing, as well as internalizing problems (primary outcomes). In addition, for parent-related outcomes the hypotheses are: 1) intervention group parents will report significantly more positive parenting practices, and coparenting support, as well as significantly fewer negative parenting practices, coparenting undermining, and parenting stress compared to control group parents (secondary outcomes); and 2) intervention group parents will report significantly more positive coping strategies with children's negative emotions and adaptive ER strategies, as well as fewer negative coping strategies with children's negative emotions and less maladaptive ER strategies in comparison with control group parents (secondary outcomes).

Additionally, the investigators aim to test potential intervention mechanisms. First, in the case of child-related outcomes, it is expected that children's use of adaptive ER strategies will mediate the intervention's effect on externalizing/internalizing problems; in a similar vein, it is hypothesized that improved social skills will mediate the intervention's effect on children's externalizing/internalizing problems. Furthermore, moderator effects of gender on adaptive emotion regulation strategies and externalizing problems will be tested.

For the parenting intervention, it is expected that program's effect on positive parenting practices and stress will be mediated by the use of positive coping strategies, parental ER and coparenting support. Also, coparenting undermining and parental reported adverse events are hypothesized to moderate the intervention's effectiveness on parenting practices, parental stress, and parent ER/coping.

DETAILED DESCRIPTION:
The first step in recruiting participants will require approaching preschool headmasters with a detailed description of the study's aims and the benefits of participating in the SEP+ intervention for both teachers and parents. All recruited schools will further inform parents of enrolled children regarding the study. Parents will be asked to provide informed consent for their children's participation in the study. Also, they will be asked to make a choice regarding their own participation to the parent training component. Afterwards, all classrooms from a particular school will be randomly assigned to either the SEP+ intervention or the wait-list control group. Data on the SEP+ effectiveness will be gathered at pre-intervention (January 2022) and at 4-months post-intervention (June 2022) for both conditions, intervention and control, respectively. Primary outcomes related to children's social-emotional skills and risk of externalizing/internalizing problems will be assessed at both baseline (T1) and immediately after the end of the intervention (T2) based on teacher and parent ratings. A similar approach will be employed for secondary outcomes. More specifically, data on self-reported parental discipline strategies, emotion regulation/coping and stress will be gathered at T1 and T2. Also, parents will be asked to fill out measures of children's social-emotional skills and externalizing/internalizing problems (primary outcomes), as well as measures related to parenting practices, parenting stress and parental ER (secondary outcomes). Both types of outcomes will be assessed at T1 and at T2, whereas parents will report about the number of adverse events only at T2. Any adverse events associated with the exposure to the classroom curriculum and/or parent training such as deterioration of child and/or parent mental health will be monitored by the research team. If such events occur, these will be reported to The Scientific Council of the Babes-Bolyai University.

As the SEP+ is comprised of multiple interventions, monitoring procedures will be employed for all components. First, regarding the implementation of the classroom curriculum, teachers will be required to fill out a self-monitoring implementation form, which will include children's attendance rates, number of implemented classroom activities, and teachers' use of intervention methods. In addition, teachers will be required to provide access to the research team to 25% filmed classroom activities. The quality of implementation for each activity by two independent raters. The teacher training will be conducted with approximately 12-15 participants in each group. Teachers will be required to participate in all 6 training sessions. Fidelity of implementation in accordance with the facilitator's manual will be conducted for half of the sessions (from sessions 2 to 5) by two independent raters based on video recordings of these sessions. Checklists will contain items describing facilitators' ability to implement specific methods of training, as well as their skills regarding group management and ways to support teachers' use of learned strategies in delivering the classroom curriculum. The parent training will also consist of 6 sessions, which will be delivered to groups of 8-10 parents. For each parent training, group fidelity checks will be conducted for 50% of the parent training sessions (sessions 2 to 5) by two independent raters based on videotaped recordings. Similar to the teacher training, facilitators will be assessed on their ability to deliver each training method according to the manual, as well as their interaction and communication skills with parents.

Approximately 30 classrooms will be recruited for the purposes of the current study. Given an expected rate of 15-30% dropout form pre- to post-intervention and that some parents might not provide consent for children to participate, the investigators estimate that the final sample will include a total of approximately 250-300 participants. A GPower a priori sample size estimation for a medium effect size, a significance level of .05 and power of .80 suggests that 41 participants are required in each group.

Data for the current study will be collected online employing Google Forms and all items will be marked mandatory to reduce the likelihood of missing data from each set of parent- and teacher-rated questionnaires. In order to handle missing data an iterative Markov chain Monte Carlo (MCMR) method will be employed.

For the purposes of the current study two types of analyses will be conducted: 1) for the effectiveness of the universal intervention (for all children in the sample), and 2) for the indicated intervention levels (children who score above the cutoff (T score > 67) on the Externalizing Problems score on the Child Behavior Checklist and the Caregiver-Teacher Report Form. For the universal intervention multi-level mixed models controlling for clustering effects will be conducted to test the intervention's effectiveness and moderator effects. Additionally, mediator effects will be tested employing multi-level meditation models in MPlus. For the indicated intervention, mixed ANOVAs will be conducted for assessing SEP+ effectiveness. Moderator and mediator effects will be assessed employing Model 1 and Model 4 from the Process add-on for Statistical Package for Social Sciences.

ELIGIBILITY:
Inclusion Criteria:

* all children for whom parental informed consent is provided
* child age between 4.5-6 years at the time of participant recruitment
* children classified at risk for externalizing problems, based on their score (cutoff T > 67) on the Externalizing Problems scale from the CBCL, and C-TRF respectively (for statistical analyses in relation to the indicated intervention)

Exclusion Criteria:

* previous child participation in a program designed to enhance social-emotional skills and/or parent participation to another parent training program
* child's age below 4.5 years or over 6 years at the time of participant recruitment
* children classified not at risk based on their score (cutoff T < 67) on the Externalizing Problems scale from the CBCL, and C-TRF respectively (for statistical analyses in relation to the indicated intervention)

Ages: 52 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 398 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Social Skills Improvement System (SSIS; Gresham & Elliott, 2002) | Change from baseline social skills at 4 months.
  The Social Skills Scale from the SSIS is a measure of children's social skills for parents and teachers. Both raters are required to assess the frequency of children's behaviors on a 4-point Likert scale ranging from 0 (never) to 3 (almost always). The scale is comprised of subscales measuring Cooperation, Communication, Assertion, Responsibility,. Empathy, Self-Control, and Engagement. Scores on each scale can be obtained by summing ratings for each item. Also, a total Social Skills score can be obtained by adding scores from each subscale.
Emotion Regulation Skills Questionnaire (ERSQ; Mirabile, 2014) | Change from baseline emotion regulation at 4 months.
  The ERSQ will be used as a measure of children's use of 13 regulatory strategies in response to negative emotions (sadness, anger, and fear) grouped into scales assessing adaptive (Self-soothing, Comfort-seeking, Support-seeking, Self-Directed Speech, Instrumental Coping, Information Gathering, Verbal Distraction, Self/Object Oriented Distraction) vs. maladaptive (Focus on Distressing Object, Venting, Aggression, Avoidance, Suppression) ER strategies. Parents and teachers rate children on their use of each ER strategy on a 4-point Likert scale ranging from 0 (never) to 3 (very much). Scores are obtained as the average scores for each regulatory strategy across the 3 emotions.
Child Behavior Checklist (CBCL; Achenbach & Rescorla, 2000) | Change from baseline externalizing/internalizing problems at 4 months.
  The CBCL is filled out by parents who are requested to respond on a 3-point Likert scale, ranging from 0 (absent) to 2 (occurs often). Responses on the Anxiety/Depression, Emotionally Reactive, Withdrawn, and Somatic Complaints will be employed for obtaining a measure of children's Internalizing Problems, whereas Aggressive Behavior and Attention Problems scores will provide a measure of Externalizing Problems. Scores for the broad-band syndrome scales are computed by adding ratings on each corresponding subscale.
Caregiver-Teacher Report Form (C-TRF; Achenbach & Rescorla, 2000) | Change from baseline externalizing/internalizing problems at 4 months.
  The C-TRF evaluates teachers' perception regarding the frequency of children's Anxiety/Depression, Emotionally Reactive, Withdrawn, Somatic Complaints, Aggressive Behaviors and Attention Problems. Responses are coded on a 3-point Likert scale, ranging from 0 (absent) to 2 (occurs often). Scores are computed by adding ratings for each type of problems and obtaining a broad-band score for either Internalizing Problems or Externalizing Problems.

SECONDARY OUTCOMES:
Parenting Young Children (PARYC; McEachern et al., 2012) | Change from baseline parental positive discipline at 4 months.
  PARYC assesses parents' use of positive discipline strategies. It comprised 21 items loading on three subscales: Supporting Positive Behavior, Limit Setting, and Proactive Parenting. Items are rated on a 7-point Likert scale, ranging from 1 (not at all) to 7 (most of the time). Scores for each scale are obtained as the average ratings for each subscale.
Parenting Scale (PS; Arnold et al., 1993) | Change from baseline over-reactivity and laxness at 4 months.
  The PS aims to assess parenting behaviors in response to children's behaviors by describing on a 7-point scale their reaction, with ratings closer to 1 suggesting more effective ways of responding, whereas ratings closer to 7 suggesting more ineffective ways of responding. Scores for the Over-reactivity and Laxness scales are computed as means.
Parental Stress Scale (PSS; Berry & Jones, 1995) | Change from baseline parental stress at 4 months.
  PSS is an 18-item measure assessing parental stress. Responses are coded on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). The Parent Stress score is obtained by summing responses to all items.
Coping with Children's Negative Emotions (CCNES; Fabes et al., 1990; Mirabile, 2015) | Change from baseline coping strategies with children's negative emotions at 4 months.
  CCNES contains 12 scenarios depicting emotion-eliciting situations for which parents are required to rate 7 possible reactions to their child's negative emotions, on a 7-point Likert scale ranging from 1 (very unlikely) to 7 (very likely). Means are obtained for each of the following scales: Distress Reactions, Punitive Reactions, Expressive Encouragement, Emotion-Focused Reactions, Problem-Focused Reactions, Minimization, and Ignoring.
Revised Parental Emotion Regulation Inventory (PERI-2; Lorber et al., 2017) | Change from baseline parental emotion regulation strategies at 4 months.
  PERI-2 contains 23 items which describe ways in which parents respond emotionally when their children misbehave. Each item is rated on a 7-point Likert scale, ranging from 1 (I never do this) to 7 (I very often do this). Means are computed for the following scales: Discipline Reappraisal, Discipline Suppression, Discipline Capitulation, and Discipline Escape.
The Coparenting Relationship Scale (CRS; Feinberg et al., 2012) | Change from baseline coparenting support and undermining at 4 months.
  The CRS measures parental perceptions about the extent to which they receive support from the partners on matters related to childrearing. Parents are requested to rate each item on a 7-point Likert scale ranging from 0 (not true of us) to 6 (very true of us). In the current study, the Coparenting Support and Coparenting Undermining will be employed.

OTHER OUTCOMES:
Adverse Events (Peterson et al., 2013) | This outcome is measured only post-intervention (approximately 4 months after the pre-intervention measure),.
  Adverse events procedures are informed by the STRONG STAR Consortium Procedure for the Monitoring of Adverse Events (a large multi-center study on Posttraumatic Stress Disorder in adults) (Peterson, Roache, Raj, & Young-McCaughan, 2013). Adverse events happening during the intervention and that are in temporal association with the participation in the study will be monitored and documented.

CONTACTS AND LOCATIONS:
Overall Officials: Catrinel A Stefan, PhD, Principal Investigator — Babes-Bolyai University
Locations (1):
- Babes-Bolyai University, Department of Psychology, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: Yes
Data collected will be anonymized, so that each participant and each intervention site will receive an identification code. IPD will be shared for each publication and will be accessible from a data repository (i.e. Open Science Framework).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Information will be available within 1 month from the time when the study's outcomes are published.
Access Criteria: Data sets pertaining to each publication will be available for all researchers. Requests concerning any other information which are not directly shared in the IPDs can be requested by email from the Principal Investigator (catrinelstefan@psychology.ro).